CLINICAL TRIAL: NCT05789940
Title: Hysteroscopy Versus Endouterine Aspiration in the Management of Trophoblastic Retention: A Prospective Randomized Multicenter Study
Brief Title: Hysteroscopy vs. Endouterine Aspiration in the Management of Trophoblastic Retention
Acronym: HARET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL22_0397
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Miscarriage
Keywords: Miscarriage; Hysteroscopy; Aspiration; Fertility; Synechiae
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Hysteroscopy (Experimental): Patients randomized to the hysteroscopy arm will receive misoprostol antibiotic prophylaxis to dilate the cervix before surgery, and anti-adhesion barrier gels will be used, according to routine procedures at each center. In case of intrauterine retention complicated by endometritis, antibiotic treatment for 48 hours (penicillin, metronidazole, fluoroquinolones or a combination of these antibiotics) will be administered according to the standard practice of each center. Evacuated retention product will be sent for pathological examination. Rh-negative women will receive prophylaxis to prevent Rh alloimmunization.
  Interventions: Procedure: hysteroscopy
- Arm B: Aspiration (Experimental): Patients randomized to the aspiration arm will receive misoprostol antibiotic prophylaxis to dilate the cervix before surgery and anti-adhesion barrier gels will be used, according to routine procedures at each center. In case of intrauterine retention complicated by endometritis, antibiotic treatment for 48 hours (penicillin, metronidazole, fluoroquinolones or a combination of these antibiotics) will be administered according to the standard practice of each center. Evacuated retention product will be sent for pathological examination. Rh-negative women will receive prophylaxis to prevent Rh alloimmunization.
  Interventions: Procedure: Aspiration

INTERVENTIONS:
Procedure: hysteroscopy — The procedure is performed by a gynecologic surgeon under general or spinal anesthesia, depending on the standard practice of the center involved, with the patient in the gynecologic position. Antibiotic prophylaxis may be administered according to the standard practice of the center. The equipment available at each center will be used for operative hysteroscopy. The use of energy is usually unnecessary and saline will be preferred. Before the operation, the appearance of the uterine cavity will be described. The selected design product will be resected from top to bottom using the surgical resector, without electrical energy, as this method is known to be the most protective of the endometrium in previous studies. Electric current should be used only as a last resort, in cases where the selected design cannot be removed without it. If there is active bleeding after the procedure, elective coagulation via the hysteroscope may be performed to stop intrauterine bleeding.
  Arms: Arm A: Hysteroscopy
Procedure: Aspiration — The aspiration will be performed by a gynecological surgeon, according to the center's standard protocol. A flexible or rigid cannula can be used. Antibiotic prophylaxis, the diameter of the cannula used, the cervical preparation required, and the use of intraoperative ultrasound guidance will be left to the discretion of the operator and the standard practice of the center. In most centers, the cervix is dilated with a Hegar dilator of up to 9 mm in size.
  Arms: Arm B: Aspiration

SUMMARY:
Introduction: Incomplete early miscarriage is defined as early miscarriage with persistent intrauterine material on ultrasound. Intrauterine retention of trophoblastic debris is not an uncommon phenomenon. These retentions may initially be asymptomatic but are often responsible for persistent metrorrhagia and endometritis. This symptomatology often accentuates the psychological distress of patients mourning the pregnancy. Incomplete miscarriages are mainly managed by the gynecological emergency department. The recommendations of the Collège National des Gynécologues et Obstétriciens Français (CNGOF) suggest as a first line of treatment: either surgical management or expectant care. The choice between the two is left to the discretion of the doctor and the patient. there are no clear recommendations as to the choice between hysteroscopy and aspiration. Within the teams, the choice is often made according to the habits and protocols of the service, according to the equipment available and the skills of the gynaecologists.

Aim: The main objective is to compare the efficacy of management by endo-uterine aspiration vs. management by hysteroscopy of trophoblastic retention after early miscarriage, at 6 weeks after surgery, by endovaginal ultrasound.

Methods: This is a prospective, multicenter, randomized, open-label, two-arms, parallel therapeutic clinical trial comparing hysteroscopy versus endouterine aspiration for the management of trophoblastic retention after spontaneous miscarriage.

Patients will be randomized (110 per arm) after verification of eligibility criteria and signature of consent, on the day of the operation:

* Arm A: 110 patients treated by operative hysteroscopy
* Arm B: 110 patients treated by endo-uterine aspiration

DETAILED DESCRIPTION:
Introduction: Incomplete early miscarriage is defined as early miscarriage with persistent intrauterine material on ultrasound. Intrauterine retention of trophoblastic debris is not an uncommon phenomenon. These retentions may initially be asymptomatic but are often responsible for persistent metrorrhagia and endometritis. This symptomatology often accentuates the psychological distress of patients mourning the pregnancy. Incomplete miscarriages are mainly managed by the gynecological emergency department. The recommendations of the Collège National des Gynécologues et Obstétriciens Français (CNGOF) suggest as a first line of treatment: either surgical management or expectant care. The choice between the two is left to the discretion of the doctor and the patient. there are no clear recommendations as to the choice between hysteroscopy and aspiration. Within the teams, the choice is often made according to the habits and protocols of the service, according to the equipment available and the skills of the gynaecologists.

Aim: The main objective is to compare the efficacy of management by endo-uterine aspiration versus management by hysteroscopy of trophoblastic retention after early miscarriage, at 6 weeks after surgery, by endovaginal ultrasound.

The secondary objectives are:

* the comparison of the rate of complications of the two techniques, during and after surgery
* the comparison of the rate of recourse to a second line surgical management between the two arms,
* the comparison of the rate of synechiae diagnosed by hysterosonography between the two techniques at 6 weeks after surgery,
* the comparison of the time to conception in the two arms during the 2 years after surgery
* the comparison of the fertility rate at 2 years after surgery in the two arms.

Methods: This is a prospective, multicenter, randomized, open-label, two-arms, parallel therapeutic clinical trial comparing hysteroscopy versus endouterine aspiration for the management of trophoblastic retention after spontaneous miscarriage.

Patients will be randomized (110 per arm) after verification of eligibility criteria and signature of consent, on the day of the operation:

* Arm A: 110 patients treated by operative hysteroscopy
* Arm B: 110 patients treated by endo-uterine aspiration Randomization will be stratified by center, age (<35 years, 35 years and over), size of trophoblastic retention (<30mm, 30mm and over) and scheduled by random size block. It will be centralized (Ennov-clinical software) and parameterized by the Unité́ de Recherche Clinique & Biostatistiques of the Montpellier University Hospital.

Statistics: The effectiveness of operative hysteroscopy is expected to be 100%, and that of aspiration 90%. To show this difference with an alpha risk of 5%, and with a power of 90%, 98 patients per arm will have to be analysed (exact binomial distribution calculation, epiR package of R implemented in biostatgv). To take into account a 10% loss of sight rate, 220 patients will be recruted.

Patients will be included in the study on the morning of the procedure, after verification of the selection criteria.

The expected number of lost to follow-up is estimated at 10%; in fact, the main criterion is evaluated relatively early (6 weeks), in patients having a desire for pregnancy and therefore relatively compliant, the rate of lost to follow-up will be a fairly low.

A flow-chart will be constructed to describe the evolution of the populations during the study. It will detail the causes of non-inclusion and the causes of loss to follow-up.

All study data will be described according to the randomization arm, in the randomized population: mean, standard deviation, median and quartiles, extrema and number of missing data for quantitative variables, numbers and percentages of each modality for qualitative data.

The clinical comparability of the randomized population and the ITT population for the primary endpoint will be assessed.

Primary analysis:

The uterine vacuity rate will be compared between the two arms in the ITT population for the primary endpoint by a Chi-square test or by a Fisher exact test if the conditions for Chi-square validity are not met. The significance level was set at 5%, two-sided.

Secondary endpoint analysis:

The rates of complications, use of second-line surgical management, synechiae, and fertility at 2 years after surgery will be compared between the two arms in their respective ITT populations, by a Chi-square test or by a Fisher's exact test if the conditions for the validity of Chi-square are not met.

The time to conception will be compared between the two arms of the randomized population by a log-rank test.

Within this family of endpoints, the alpha risk will be controlled by a Hochberg procedure.

Visit 1: Pre-operative consultation between 1 and 21 days before the operation

* Clinical examination performed as part of routine care: measurement of blood pressure and pulse, temperature, speculum examination to ensure the absence of significant bleeding indicating emergency surgical management.
* Diagnosis of trophoblastic retention by endovaginal ultrasound

At the end of the consultation:

* Verification of eligibility criteria
* Oral information on the study and information leaflet given to the patient
* Collection of informed and written consent after a reflection period
* Collection of the following data:
* Demographic data
* History, smoking habits and concomitant treatments
* Pregnancy data leading to the current miscarriage
* Results of pelvic ultrasound

Intervention (D0):

* Verification of eligibility criteria and randomization on the morning of the procedure
* Surgical management of trophoblastic retention by operative hysteroscopy (Arm A) or endo-uterine aspiration (Arm B)
* Collection of adverse events during the operation and before the patient is discharged

Visit 2: Consultation at 6 weeks after surgery +/- 7 days

This consultation will be performed by an investigator trained in pelvic ultrasound and hysterosonography, blinded to the allocated procedure:

* Plasma HCG measurement before hysterosonography to ensure that there is no current pregnancy
* Endovaginal ultrasound to check uterine vacuity
* Hysterosonography for the diagnosis of uterine synechia
* Collection of complications and adverse events after surgery

Visit 3: Telephone consultation at 6 months +/- 15 days after surgery

Carried out by the clinical research associate (CRA):

* Evaluation of fertility by questionnaire
* Evaluation of the time to conception if pregnancy in progress A letter will be sent to the patient if she cannot be reached by phone (questionnaire + return envelope)

Visit 4: Telephone consultation at 12 months +/- 1 month after surgery

Carried out by the CRA:

* Evaluation of fertility by questionnaire.
* Evaluation of the time to conception if pregnancy in progress. A letter will be sent to the patient if she cannot be reached by phone (questionnaire + return envelope)

Visit 5: Telephone consultation at 24 months (+/- 2 months) after surgery

Carried out by the CRA:

* Evaluation of fertility by questionnaire
* Evaluation of the time to conception if pregnancy in progress A letter will be sent to the patient if she cannot be reached by phone (questionnaire + return envelope). The patients will be followed until a pregnancy is obtained with a term greater than or equal to 24 weeks of amenorrhea or over a maximum period of 26 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Management for trophoblastic retention after early spontaneous miscarriage (<14 weeks of amenorrhea)
* Diagnosis of intrauterine trophoblastic retention by endovaginal pelvic ultrasound
* Shared decision for surgical management
* Current pregnancy desire

Exclusion Criteria:

* Known uterine malformation
* Patient who has received surgical treatment for current intrauterine retention
* Trophoblastic retention after elective termination, late miscarriage and postpartum
* Patient with an intrauterine device (IUD)
* Pregnancy obtained by medically assisted procreation
* Indication for emergency surgical management for haemostatic purposes
* Failure to obtain free, informed and written consent after a period of reflection
* Person not affiliated or beneficiary of a national health insurance system
* Person protected by law, under guardianship or curatorship
* Person participating in other interventional research involving the human person

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Uterine vacuity | 6 weeks after surgery
  Uterine vacuity will be determined by endovaginal pelvic ultrasound. The endovaginal pelvic ultrasound will be performed by an investigator blinded to the patient's group, in order to minimize bias. It will be performed according to a standard pelvic ultrasound technique: a sagittal section and a transverse section passing through the widest part of the uterine body. Uterine vacuity will be defined by a thickness of the mucosa on a sagittal section of 15 mm or less and the absence of a heterogeneous intrauterine mass

SECONDARY OUTCOMES:
Difference between the two arms in complication rates | During surgery and 6 weeks after surgery
  Complications will be described according to clavien-dindo classification
Difference between the two arms in the rate of second line surgical management | During surgery
  The rate of second line surgical management will be described
Difference between the two arms in synechia rates | 6 weeks after surgery
  Presence of synechia will be assessed by hysterosonography
Difference between the two arms in mean time to conception | 6, 12 and 24 months after surgery
  Patients will be contacted by phone at 6, 12 and 24 months after the surgery to ask if they have been pregnant et evaluate the time of conception
Difference between the two arms in pregnancy rates | 6, 12 and 24 months after surgery
  Patients will be contacted by phone at 6, 12 and 24 months after the surgery to assess their fertility

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, MD, Study Director — CHU de Montpellier
Locations (4):
- France (4):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Nice - Hôpital Archet II, Nice
  - CHU de Nîmes - Hôpital Carémeau, Nîmes

IPD SHARING:
Plan to Share IPD: No